CLINICAL TRIAL: NCT05173415
Title: MALLORCA - Trial (Surgical MArker LocaLisation OR Clip and Wire Application for Targeted Axillary Dissection in Node Positive Breast Cancer Patients) A Prospective, Randomized Multi-centre Trial.
Brief Title: Marker Technique Comparison in Targeted Axillary Dissection
Acronym: MALLORCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Constanze Elfgen (Other)
Responsible Party: Sponsor-Investigator, Constanze Elfgen, Study Principal Investigator, Brust-Zentrum AG
Organization: Brust-Zentrum AG (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 021-013772
Record Dates: First submitted 2021-10-28; First posted 2021-12-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: A prospective, randomized multi-centre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirius Pintution Group (Experimental): Patients who are randomized for the Pintution Clip will receive a preoperative ultrasound-guided marking in the axillary lymph nodes that indicate for surgical removal. Surgical procedure is standardized with a handheld probe leading intraoperatively to the marked lymph node and its excision. Successful detection, time of the procedure (beginning of localization intervention to completed lymph node excision), and intra- and postoperative complication rate will be measured. Intra- and postoperative complications are adverse events during the surgery or within 48 hours after the surgery.
  Interventions: Device: Sirius Pintution
- HydroMARK(C) Clip Group (Active Comparator): Patients who are randomized for the standard clip will receive a preoperative ultrasound-guided marking with HydroMark® Clip in the axillary lymph node that indicate for surgical removal. Surgical procedure is standardized with intraoperative ultrasound-guided wire-localization of the clip and lymph node excision. Successful detection, time of the procedure (beginning of localization intervention to completed lymph node excision), and intra- and postoperative complication rate will be measured. Intra- and postoperative complications are adverse events during the surgery or within 48 hours after the surgery.
  Interventions: Device: HydroMARK (C) Clip

INTERVENTIONS:
Device: Sirius Pintution — The intervention studies a metal Clip (Sirius Pintution) to localize axillary lymph nodes during TAD. Intraoperative localization of the lymph node will be conducted using a hand-held probe identifying the clip.
  Arms: Sirius Pintution Group
Device: HydroMARK (C) Clip — The control intervention is a metal clip (HydroMARK© Clip), which will be localized and extracted during the tailoring surgery. Intraoperative Ultrasound is used to localize the clip. This method is considered as standard practice today.
  Arms: HydroMARK(C) Clip Group

SUMMARY:
Comparison of two methods (Magnetic Marker and standard metal clip) used for localisation and extraction of lymph nodes in Targeted Axillary Dissection (TAD) in patients with breast cancer.This Project will investigate and compare the duration of intervention, detection rate and safety.

The participants will be randomized into two groups of equal size.

DETAILED DESCRIPTION:
This Project will investigate and compare the duration of intervention, detection rate and safety of two methods (Magnetic Sirius Pintuition Marker and standard metal clip) used for the localisation and extraction of lymph nodes in Targeted Axillary Dissection (TAD).

The participants will be randomized into two groups of equal size. The groups differ in terms of the method used to mark the lymph nodes prior to TAD. One group will receive a metal clip (HydroMARK© Clip), which will be localized and extracted during the tailoring surgery. Intraoperative Ultrasound is used to localize the clip. This method is considered as standard practice today.

The second group will receive Metal Clip (Sirius Pintuition) to localize axillary lymph nodes during TAD. Intraoperative localization of the lymph node will be conducted using a hand-held probe.

Successful localization of the lymph node, duration of the intervention (beginning of the localization until successful extraction) and adverse effects will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Indication: Patients undergoing lymph node marking before targeted axillary dissection due to suspicious lymph nodes or confirmed lymph node metastasis in breast cancer patients
* Female participants ≥ 18 years of age
* The subject was informed about the project and gave her written informed consent to use her data and samples for this project.
* BMI < 30
* Indication for neoadjuvant chemotherapy

Exclusion Criteria:

* Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
To compare clinical manageability, efficacy, safety, and sufficiency of two lymph node marking systems (HydroMark Clip versus Sirius Pintuition) | 6 months
  The primary outcome is the efficacy of both methods for lymph node marking. Efficacy is defined as performance time during the surgery from skin incision (either with hooked wire or scalpel) until the complete excision of the marked lymph node. Time is measured in minutes. Manageability includes process performance of the marker insertion (questionnaire for the study physician: "did you experience problems or barriers in inserting the marker?"; "if yes, what kind of?"). Safety is also observed via the questionnaire ("did your patient experience adverse events? bleeding, seroma, (...), other?"). This is also true for sufficiency ("Did you acieve a successful lymph node marking?"; "Have you been able to localize the marker during the surgery or has it been dislocated?"; "Did you manage to remove the marked lymph node including the marker").

SECONDARY OUTCOMES:
Failure rate (unsuccessful localisation of the marked lymph node) | 6 months
  As a secondary outcome, the failure rate (unsuccessful localisation of the marked lymph node) will be measured. As the failure rate is supposed to be low in general, this topic is not the focus of our study.
Incidence of complications of both methods used for lymph node marking. | 6 months
  This outcome measures the safety of both methods during the implantation of the randomised marker, excision surgery of the lymph node and postoperative period.
Adverse events | 6 months
  This outcome assesses adverse events caused by either lymph node marker during implantation and excision of the marker and within the postoperative period.
Satisfaction of the performing Surgeon concerning the handling of the marking technique documented in the Case Report Form. | 6 months
  This outcome measures the satisfaction of the performing surgeon concerning the handling of the lymph node marking technique during implantation and excision surgery.

OTHER OUTCOMES:
Incidence of intraoperative complications and postoperative adverse events. | 6 months
  The safety outcome variables include allergic reactions, bleeding, bruising, dislocation, pain, scar, and very rare events such as lymphedema or neurologic damages.

CONTACTS AND LOCATIONS:
Overall Officials: Constanze Elfgen, Dr.med., Principal Investigator — Brust-Zentrum AG
Locations (4):
- Switzerland (4):
  - Brustzentrum Kantonsspital Baden, Baden, Canton of Aargau
  - Brustzentrum Bern Biel, Bern
  - Brustzentrum Ostschweiz, Sankt Gallen
  - Brust-Zentrum Zürich AG, Zurich

IPD SHARING:
Plan to Share IPD: No